CLINICAL TRIAL: NCT03943966
Title: In-vivo Thrombus Imaging With 18F-GP1, a Novel Platelet PET Radiotracer
Acronym: iThrombus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: British Heart Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: AC18071
Record Dates: First submitted 2019-04-22; First posted 2019-05-09 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: Thrombosis; Atherothrombosis; Myocardial Infarction; STEMI; NSTEMI - Non-ST Segment Elevation MI; DVT; Pulmonary Embolism; Stroke; Transient Ischemic Attack; Prosthetic Valve Thrombosis; PET
MeSH Terms: conditions — Thrombosis; Myocardial Infarction; ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction; Pulmonary Embolism; Stroke; Ischemic Attack, Transient

STUDY DESIGN:
Intervention Model Description: Single centre prospective pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Myocardial Infarction (Experimental)
  Interventions: Diagnostic Test: 18F-GP1 PET CT
- Stable coronary disease with intracoronary stent insertion (Active Comparator)
  Interventions: Diagnostic Test: 18F-GP1 PET CT
- Deep vein thrombosis and Pulmonary embolus (Active Comparator)
  Interventions: Diagnostic Test: 18F-GP1 PET CT
- Surgical and Transcatheter Aortic valve replacement (Active Comparator)
  Interventions: Diagnostic Test: 18F-GP1 PET CT
- Transient ischaemic attack and stroke (Active Comparator)
  Interventions: Diagnostic Test: 18F-GP1 PET CT

INTERVENTIONS:
Diagnostic Test: 18F-GP1 PET CT — PET CT scan using platelet radiotracer 18F-GP1

SUMMARY:
To date, the investigators have successfully employed a radiotracer (18F-sodium fluoride) as a marker of necrotic inflammation in human atherosclerosis. The investigators aim to further the mechanistic understanding of atherothrombosis by studying the activation of glycoprotein IIb/IIIa receptors in cardiovascular thrombus using the novel platelet radiotracer (18F-GP1). Binding of 18F-GP1 to activated platelets in venous and arterial thrombi has already been demonstrated in pre-clinical studies and a phase 1 trial in man. If successful, this study would define the role of the glycoprotein IIb/IIIa receptor within in vivo thrombosis across a range of cardiovascular diseases.

DETAILED DESCRIPTION:
Cardiovascular thrombotic conditions were estimated to account for 1 in 4 deaths worldwide in 2010 and are the leading cause of global mortality. Divided into arterial and venous thromboses, ischaemic heart disease and ischemic stroke comprise the major arterial thromboses and deep-vein thrombosis and pulmonary embolism comprise the major venous thromboses. Although both arterial and venous thrombi differ in both aetiology and pathophysiology, many commonalities remain.

Thrombosis begins with damage to the vascular wall. Physiological haemostasis is triggered when underlying collagen is exposed to circulating platelets which bind directly to collagen with collagen-specific glycoprotein surface receptors. After an initial signalling cascade involving release of platelet binder von Willebrand Factor, platelets become activated which allows adherence to the site of injury. Following activation, phospholipase A2 modifies the integrin membrane glycoprotein IIb/IIIa (GP IIb/IIIa) increasing platelet ability to bind fibrinogen. The activated platelets then change shape from spherical to stellate, and the fibrinogen cross-links with glycoprotein IIb/IIIa aiding aggregation of more platelets and completing primary haemostasis. Secondary haemostasis involves activation of the coagulation cascade through extrinsic and intrinsic pathways and ends with cross linked fibrin deposition and a mature thrombus.

The haemostatic process is fluid and dynamic with the expression of activated membrane proteins and coagulation factors changing throughout. Platelet expression of GP IIb/IIIa falls as a thrombus matures hence why it is a pharmacological target for antithrombotic therapies. The investigators aim to explore the expression and distribution of GP IIb/IIIa receptors in a range of thrombotic conditions listed below spanning across both arterial and venous systems. Improving understanding of how clinical presentation relates to platelet activation over a range of conditions is crucially important when deciding appropriate anti-thrombotic regimes.

1.2.1 Coronary Heart Disease and Myocardial Infarction Coronary heart disease is the leading cause of death worldwide and is responsible for 17.5 million or 46% of all non-communicable deaths in 2012. The majority of the cardiovascular morbidity and mortality is attributable to coronary atherosclerosis and thrombosis. Atherosclerosis is the central process by which the heart arteries narrow and harden due to the deposition of fatty plaques within the artery wall. This process can result in damage to the lining of the artery which can cause a thrombus (clot) to form within the artery which can partially or completely occlude the flow of blood to the heart muscle thereby precipitating myocardial infarction. This is the commonest form of a heart attack and responsible for a large proportion of sudden cardiac deaths. Thrombus in myocardial infarction is classically thought to be composed of predominantly platelets. However, recent research has shown that 56% of thrombus in MI is composed of fibrin with only 17% platelets. Ischaemic time correlated positively with thrombus fibrin content and negatively with thrombus platelet component. This illustrates the dynamic interaction between platelets and fibrin over time.

1.2.2 Bioprosthetic heart valve thrombosis Bioprosthetic valve thrombosis is an increasingly recognised complication of valve replacement. Patient risks include early prosthesis failure requiring redo operation plus stroke or other systemic embolism. A meta-analysis has estimated the incidence of bioprosthetic thrombosis to be 0.03 per 100 patient years with the risk of embolism being highest in the first 3 months post implantation. The composition of prosthetic valve thrombosis varies depending on valve type and time from insertion. Interestingly in the MISTRAL-C randomised controlled trial, 50% of acute thromboembolic events within 3 days of transcatheter aortic valve insertion were platelet-fibrin thrombus, not calcific debris from the aortic root. Thromboembolism was less common in those on anticoagulant rather than antithrombotic treatment suggesting a fibrin predominance. Similar results were found in a large registry of over 25,000 patients undergoing surgical bioprosthetic valve insertion. Warfarin plus aspirin was more effective than aspirin alone in preventing thromboembolic events and death.

1.2.3 Venous thromboembolic disease Pulmonary embolism is a common cardiovascular condition with a high morbidity and mortality. Embolisation of a venous thrombosis from the deep veins of the lower limbs or pelvis is the aetiology in more than 90% events. Thrombus formation is triggered by intravascular activation of coagulation and thrombin-mediated intraluminal fibrin deposition. Red blood cells (RBCs) are thought to be incorporated into venous thrombi via passive trapping in the growing fibrin network, culminating in the production of a RBC and fibrin rich venous thrombus. Treatment for both DVT and PE reduces mortality and secondary prophylaxis with anticoagulation is effective at preventing further events. The clinically most frequently applied imaging test for visualisation of suspected PE is CT pulmonary angiography (CTPA). For DVT, a range of imaging modalities can be used (US, CT or MR) with ultrasound the most common first line investigation.

1.2.4 Stroke and Transient Ischaemic Attack (TIA) Stroke and TIA are leading causes of preventable death and morbidity worldwide. Thrombus composition is thought to depend on source (cardiac chamber or head or neck artery) and time from event. Fibrin-dominant thrombus is likely to be more refractory to thrombolytic drugs as is the presence of chronic histopathologic features in clots such as endothelialisation and calcification. Diagnosis is based on clinical presentation followed by CT or MRI of the brain with US or MR assessment of carotid stenosis performed thereafter to ascertain future event risk.

1.2.5 COVID-19 The COVID-19 pandemic has resulted in major mortality and morbidity. Consistent clinical concerns have been raised in published literature, news outlets and social media regarding thromboembolic events affecting the microvasculature as well as large vessels. This has received widespread attention and led to the reported use of prophylactic or therapeutic anticoagulation regimes, or even fibrinolysis, outwith standard protocols and indications in the absence of firm evidence of clinical benefit, such is the concern. Given its sensitivity for detecting activated platelets, which our pilot data has suggested may be superior to other imaging modalities in some settings, 18F-GP1 PET-CT may offer a suitable method to examine the posited association between COVID-19 and thromboembolic disease.

1.3 Understanding Platelet Biology As platelet aggregation is a major component of both arterial and venous thrombi, the investigators propose to explore whether a radiolabelled ligand (18F-GP1) of the glycoprotein IIb/IIIa (GPIIb/IIIa) receptor can detect activated platelets on thrombus. GPIIb/IIIa receptors mediate platelet adherence and aggregation. They are expressed in greater numbers and assume a more ligand binding conformation on activation which binds protein ligands including von Willebrand factor and Fibrinogen. This allows for platelet bridging and aggregation. Accordingly, they represent an attractive target for acute thrombus imaging. We hope to identify activated platelets in the five groups presented above. Identification of activated platelets in all conditions will further enhance our understanding of the role of this receptor in both arterial and venous thrombosis and how anti-thrombotic therapy influences expression.

1.4 Glycoprotein IIb/IIIa inhibition Three intravenous platelet glycoprotein (GP) IIb/IIIa inhibitors have been studied extensively and are available for clinical use: abciximab, tirofiban, and eptifibatide. Abciximab is a monoclonal antibody directed against the receptor, while tirofiban and eptifibatide are high affinity non-antibody receptor inhibitors.

Antiplatelet therapy with intravenous GP IIb/IIIa inhibitors has been evaluated in patients with acute coronary syndrome (ACS) and in those undergoing intracoronary stent implantation and stroke but not DVT/PE or prosthetic valve implantation.

Meta-analyses have evaluated the use of intravenous glycoprotein (GP) IIb/IIIa inhibitors in a variety of settings related to coronary disease. The impact of the intravenous GP IIb/IIIa inhibitors on clinical outcomes was assessed in a pooled analysis of 21 trials involving various groups of patients with ischemic heart disease. The GP IIb/IIIa inhibitor reduced the combined end point of death, nonfatal myocardial infarction (MI), or urgent revascularization at 30 days in the following groups of patients:

* Those undergoing a percutaneous coronary intervention (PCI)
* Those with non-ST elevation myocardial infarction (NSTEMI)
* Those with an ST elevation MI (STEMI) treated with percutaneous transluminal coronary angioplasty (PTCA) However, these trials were performed largely before the routine use drug eluting stents and dual oral antiplatelet therapy with aspirin and a platelet P2Y12 receptor blocker. In summary, the role of P2Y12 inhibitors has decreased the role of GP IIb/IIIa therapy in coronary heart disease, although it continues to be important in some subgroups of patients. We aim to explore the expression of activated platelets within both stable and unstable coronary disease and how PCI and use of anti-thrombotic drugs (P2Y12 and GPIIb/IIIa inhibitors) mediate expression.

In stroke disease, a single randomised controlled trial (SaTIS) performed in moderate ischaemic stroke demonstrated a significant reduction in mortality at 5 months with tirofiban when compared to placebo. Importantly there was no difference in major haemorrhage.The investigators aim to explore the expression of GPIIb/IIIa in stroke and TIA and explore how it may differ in the embolised thrombus when compared with the culprit plaque.

Efficacy of GPIIb/IIIa inhibition in recent bioprosthetic valve insertion and DVT/PE is unknown. We aim to explore activated platelet expression in both conditions to gain insight as to whether GPIIb/IIIa inhibition may be a potentially useful treatment.

1.5 Background of 18F-GP1 GP1 is a ligand of the fiban class of molecule which has a high affinity for the glycoprotein IIb/IIIa receptor; highly expressed on activated platelets. It is an excellent target for imaging arterial thrombi with a large activated platelet component. After a 2 step radiofluorination subsequent purification process 18F-GP1 can be used for PET imaging.

18F-GP1 has undergone pre-clinical and phase 1 clinical evaluation demonstrating a high affinity to GPIIb/IIIa, the key receptor for platelet aggregation. It binds in a stable and specific manner to in vivo arterial, venous and intracardiac human thrombus. Binding is crucially not altered by anticoagulation therapy (aspirin and heparin).

In the recent phase 1 study 18F-GP1 demonstrated a high detection rate of thromboembolic foci in 20 patients with recently formed deep vein thrombi (DVT) and pulmonary thromboemboli. The tracer also performed favourably with regards to its metabolism, pharmacokinetic and dosimetry profile. There were no significant adverse events in any of the 20 recruited participants.

1.6 Study Aims

We aim to examine the expression of the glycoprotein IIb/IIIa receptor in:

1. Intracoronary thrombus following spontaneous myocardial infarction
2. Intracoronary thrombus following routine stent insertion.
3. Bioprosthetic heart valve thrombosis (surgical or transcatheter valves).
4. Venous thromboembolic disease in those with recently confirmed deep vein thrombosis and pulmonary embolism.
5. Carotid and cerebral thrombus in those with stroke and TIA. This would enhance our understanding of the incidence, consequences and natural history of platelet activation within cardiovascular thrombosis.

1.7 Research Hypothesis

GPIIb/IIIa receptor expression is varied by thrombotic condition including venous (DVT/PE) versus arterial (MI/stroke), in situ (MI) versus embolic (stroke, PE) and prosthetic material (stents and valves) versus diseased native tissue (MI, stroke, DVT/PE).

1.8 Rationale for Study To date, the investigators have successfully employed a radiotracer (18F-sodium fluoride) as a marker of necrotic inflammation in human atherosclerosis. Binding of 18F-GP1 to activated platelets in venous and arterial thrombi has already been demonstrated in pre-clinical studies and a phase 1 trial in man. If successful, this study would define the role of the glycoprotein IIb/IIIa receptor within in vivo thrombosis across a range of cardiovascular diseases.

ELIGIBILITY:
4.2 Myocardial infarction group inclusion/exclusion criteria 4.2.1 Myocardial infarction Inclusion criteria

* Male or females over the age of 40 with recent (within 7 days) type 1 myocardial infarction (21) awaiting or have undergone inpatient coronary angiography, or with suspected myocardial infarction in the context of confirmed COVID-19 requiring hospital admission.
* Provision of informed consent prior to any study specific procedures

4.2.2 Myocardial infarction Exclusion Criteria Subjects should not enter the study if any of the following criteria are fulfilled

* Inability or unwilling to give informed consent.
* Unable to tolerate the supine position
* Impaired renal function with eGFR of <30 mL/min/1.73m2
* Allergy to iodinated contrast
* Severe or significant comorbidity
* Women who are pregnant or breastfeeding

4.3 Stable CAD inclusion/exclusion criteria

4.3.1 Stable CAD inclusion criteria

* Male or females over the age of 40 with stable coronary artery disease who have undergone a recent (<30 days) coronary angiogram + PCI
* Provision of informed consent prior to any study specific procedures

4.3.2 Stable coronary disease exclusion criteria

* Myocardial infarction less than 3 months ago
* Inability or unwilling to give informed consent.
* Unable to tolerate the supine position
* Allergy to iodinated contrast
* Impaired renal function with eGFR of <30 mL/min/1.73m2
* Severe or significant comorbidity
* Women who are pregnant or breastfeeding

4.4 Bioprosthetic heart valve inclusion/exclusion criteria

4.4.1 Bioprosthetic aortic valve inclusion criteria

* Ability to give informed consent
* Males or females over 40 years of age with recent (up to 6±4 weeks) surgical bioprosthetic heart valve replacement (SAVR or SMVR) or transcatheter bioprosthetic heart valve insertion (TAVI or TMVR).

4.4.2 Bioprosthetic heart valve exclusion criteria

* Inability to give informed consent
* Pregnancy
* Breastfeeding
* Claustrophobia
* Allergy to iodinated contrast
* Liver failure
* Chronic kidney disease (with estimated glomerular filtration rate <30 mL/min)
* Paget's disease
* Metastatic malignancy
* Inability to tolerate the supine position
* Women who are pregnant or breastfeeding

4.5 DVT/PE inclusion/exclusion criteria 4.5.1 DVT/PE inclusion criteria

* Male or females over the age of 40 with recently confirmed (<30 days) DVT on ultrasound or PE on CTPA as per ESC diagnostic guidelines (22), or with suspected DVT or PE in the context of confirmed COVID-19 requiring hospital admission
* Provision of informed consent prior to any study specific procedures

4.5.2 DVT/PE exclusion criteria

* Inability or unwilling to give informed consent.
* Unable to tolerate the supine position
* Impaired renal function with eGFR of <30 mL/min/1.73m2
* Allergy to iodinated contrast
* Contraindication to iodinated contrast agents
* Severe of significant comorbidity
* Women who are pregnant or breastfeeding
* Contra-indication to Magnetic Resonance imaging in the 6 patients offered PET MR scanning.

4.6 Stroke and TIA inclusion/exclusion criteria

4.6.1 Stroke and TIA inclusion criteria

* Male or females over the age of 40 with recently diagnosed stroke or TIA as per diagnostic criteria of the American Heart and Stroke Association guidelines (23), with or without COVID-19.
* Provision of informed consent prior to any study specific procedures

4.6.2 Stroke and TIA exclusion criteria

* Inability or unwilling to give informed consent.
* Unable to tolerate the supine position
* Impaired renal function with eGFR of <30 mL/min/1.73m2
* Allergy to iodinated contrast
* Contraindication to iodinated contrast agents
* Severe of significant comorbidity
* Women who are pregnant or breastfeeding

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2019-11-11 (Actual); Primary Completion 2021-07-02 (Actual); Study Completion 2021-10-13 (Actual)

PRIMARY OUTCOMES:
Ratio of 18F-GP1 standardised uptake values (SUV's) in thrombus compared with the SUVs recorded in the blood pool. | 6 months from end of recruitment
  Expression of the glycoprotein IIb/IIIa receptor (assessed by SUV) within thrombus in the arterial and venous circulation.

SECONDARY OUTCOMES:
Ratio of 18F-GP1 standardised uptake values (SUV's) in thrombus formed in each of the 5 disease states. | 6 months from end of recruitment
  Expression of the glycoprotein IIb/IIIa receptor (assessed by SUV) within thrombus in the arterial and venous circulation in all 5 disease states

CONTACTS AND LOCATIONS:
Locations (1):
- University of Edinburgh, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wendelboe AM, Raskob GE. Global Burden of Thrombosis: Epidemiologic Aspects. Circ Res. 2016 Apr 29;118(9):1340-7. doi: 10.1161/CIRCRESAHA.115.306841. PMID 27126645
- [Background] Organisation WH. Cardiovascular diseases 2018 [Available from: www.who.int/cardiovascular_diseases/en/
- [Background] Silvain J, Collet JP, Nagaswami C, Beygui F, Edmondson KE, Bellemain-Appaix A, Cayla G, Pena A, Brugier D, Barthelemy O, Montalescot G, Weisel JW. Composition of coronary thrombus in acute myocardial infarction. J Am Coll Cardiol. 2011 Mar 22;57(12):1359-67. doi: 10.1016/j.jacc.2010.09.077. PMID 21414532
- [Background] Puvimanasinghe JP, Steyerberg EW, Takkenberg JJ, Eijkemans MJ, van Herwerden LA, Bogers AJ, Habbema JD. Prognosis after aortic valve replacement with a bioprosthesis: predictions based on meta-analysis and microsimulation. Circulation. 2001 Mar 20;103(11):1535-41. doi: 10.1161/01.cir.103.11.1535. PMID 11257081
- [Background] Heras M, Chesebro JH, Fuster V, Penny WJ, Grill DE, Bailey KR, Danielson GK, Orszulak TA, Pluth JR, Puga FJ, et al. High risk of thromboemboli early after bioprosthetic cardiac valve replacement. J Am Coll Cardiol. 1995 Apr;25(5):1111-9. doi: 10.1016/0735-1097(94)00563-6. PMID 7897124
- [Background] Van Mieghem NM, van Gils L, Ahmad H, van Kesteren F, van der Werf HW, Brueren G, Storm M, Lenzen M, Daemen J, van den Heuvel AF, Tonino P, Baan J, Koudstaal PJ, Schipper ME, van der Lugt A, de Jaegere PP. Filter-based cerebral embolic protection with transcatheter aortic valve implantation: the randomised MISTRAL-C trial. EuroIntervention. 2016 Jul 20;12(4):499-507. doi: 10.4244/EIJV12I4A84. PMID 27436602
- [Background] Brennan JM, Edwards FH, Zhao Y, O'Brien S, Booth ME, Dokholyan RS, Douglas PS, Peterson ED; DEcIDE AVR Research Team. Early anticoagulation of bioprosthetic aortic valves in older patients: results from the Society of Thoracic Surgeons Adult Cardiac Surgery National Database. J Am Coll Cardiol. 2012 Sep 11;60(11):971-7. doi: 10.1016/j.jacc.2012.05.029. Epub 2012 Aug 22. PMID 22921973
- [Background] Heit JA, Spencer FA, White RH. The epidemiology of venous thromboembolism. J Thromb Thrombolysis. 2016 Jan;41(1):3-14. doi: 10.1007/s11239-015-1311-6. PMID 26780736
- [Background] Sevitt S. The structure and growth of valve-pocket thrombi in femoral veins. J Clin Pathol. 1974 Jul;27(7):517-28. doi: 10.1136/jcp.27.7.517. PMID 4138834
- [Background] Darbousset R, Thomas GM, Mezouar S, Frere C, Bonier R, Mackman N, Renne T, Dignat-George F, Dubois C, Panicot-Dubois L. Tissue factor-positive neutrophils bind to injured endothelial wall and initiate thrombus formation. Blood. 2012 Sep 6;120(10):2133-43. doi: 10.1182/blood-2012-06-437772. Epub 2012 Jul 26. PMID 22837532
- [Background] Wells PS, Ihaddadene R, Reilly A, Forgie MA. Diagnosis of Venous Thromboembolism: 20 Years of Progress. Ann Intern Med. 2018 Jan 16;168(2):131-140. doi: 10.7326/M17-0291. Epub 2018 Jan 9. PMID 29310137
- [Background] Feigin VL, Forouzanfar MH, Krishnamurthi R, Mensah GA, Connor M, Bennett DA, Moran AE, Sacco RL, Anderson L, Truelsen T, O'Donnell M, Venketasubramanian N, Barker-Collo S, Lawes CM, Wang W, Shinohara Y, Witt E, Ezzati M, Naghavi M, Murray C; Global Burden of Diseases, Injuries, and Risk Factors Study 2010 (GBD 2010) and the GBD Stroke Experts Group. Global and regional burden of stroke during 1990-2010: findings from the Global Burden of Disease Study 2010. Lancet. 2014 Jan 18;383(9913):245-54. doi: 10.1016/s0140-6736(13)61953-4. PMID 24449944
- [Background] Singh P, Kaur R, Kaur A. Clot composition and treatment approach to acute ischemic stroke: The road so far. Ann Indian Acad Neurol. 2013 Oct;16(4):494-7. doi: 10.4103/0972-2327.120433. PMID 24339566
- [Background] Dobrucki LW, Sinusas AJ. PET and SPECT in cardiovascular molecular imaging. Nat Rev Cardiol. 2010 Jan;7(1):38-47. doi: 10.1038/nrcardio.2009.201. Epub 2009 Nov 24. PMID 19935740
- [Background] Sabatine MS, Jang IK. The use of glycoprotein IIb/IIIa inhibitors in patients with coronary artery disease. Am J Med. 2000 Aug 15;109(3):224-37. doi: 10.1016/s0002-9343(00)00474-5. PMID 10974186
- [Background] Siebler M, Hennerici MG, Schneider D, von Reutern GM, Seitz RJ, Rother J, Witte OW, Hamann G, Junghans U, Villringer A, Fiebach JB. Safety of Tirofiban in acute Ischemic Stroke: the SaTIS trial. Stroke. 2011 Sep;42(9):2388-92. doi: 10.1161/STROKEAHA.110.599662. Epub 2011 Aug 18. PMID 21852609
- [Background] Nurden AT. Inherited abnormalities of platelets. Thromb Haemost. 1999 Aug;82(2):468-80. No abstract available. PMID 10605738
- [Background] Lohrke J, Siebeneicher H, Berger M, Reinhardt M, Berndt M, Mueller A, Zerna M, Koglin N, Oden F, Bauser M, Friebe M, Dinkelborg LM, Huetter J, Stephens AW. 18F-GP1, a Novel PET Tracer Designed for High-Sensitivity, Low-Background Detection of Thrombi. J Nucl Med. 2017 Jul;58(7):1094-1099. doi: 10.2967/jnumed.116.188896. Epub 2017 Mar 16. PMID 28302764
- [Background] Joshi NV, Vesey AT, Williams MC, Shah AS, Calvert PA, Craighead FH, Yeoh SE, Wallace W, Salter D, Fletcher AM, van Beek EJ, Flapan AD, Uren NG, Behan MW, Cruden NL, Mills NL, Fox KA, Rudd JH, Dweck MR, Newby DE. 18F-fluoride positron emission tomography for identification of ruptured and high-risk coronary atherosclerotic plaques: a prospective clinical trial. Lancet. 2014 Feb 22;383(9918):705-13. doi: 10.1016/S0140-6736(13)61754-7. Epub 2013 Nov 11. PMID 24224999
- [Background] Dweck MR, Chow MW, Joshi NV, Williams MC, Jones C, Fletcher AM, Richardson H, White A, McKillop G, van Beek EJ, Boon NA, Rudd JH, Newby DE. Coronary arterial 18F-sodium fluoride uptake: a novel marker of plaque biology. J Am Coll Cardiol. 2012 Apr 24;59(17):1539-48. doi: 10.1016/j.jacc.2011.12.037. PMID 22516444
- [Background] Thygesen K, Alpert JS, Jaffe AS, Simoons ML, Chaitman BR, White HD; Writing Group on behalf of the Joint ESC/ACCF/AHA/WHF Task Force for the Universal Definition of Myocardial Infarction. Third universal definition of myocardial infarction. Glob Heart. 2012 Dec;7(4):275-95. doi: 10.1016/j.gheart.2012.08.001. Epub 2012 Sep 26. No abstract available. PMID 25689940
- [Background] Konstantinides SV, Torbicki A, Agnelli G, Danchin N, Fitzmaurice D, Galie N, Gibbs JS, Huisman MV, Humbert M, Kucher N, Lang I, Lankeit M, Lekakis J, Maack C, Mayer E, Meneveau N, Perrier A, Pruszczyk P, Rasmussen LH, Schindler TH, Svitil P, Vonk Noordegraaf A, Zamorano JL, Zompatori M; Task Force for the Diagnosis and Management of Acute Pulmonary Embolism of the European Society of Cardiology (ESC). 2014 ESC guidelines on the diagnosis and management of acute pulmonary embolism. Eur Heart J. 2014 Nov 14;35(43):3033-69, 3069a-3069k. doi: 10.1093/eurheartj/ehu283. Epub 2014 Aug 29. No abstract available. PMID 25173341
- [Background] Sacco RL, Kasner SE, Broderick JP, Caplan LR, Connors JJ, Culebras A, Elkind MS, George MG, Hamdan AD, Higashida RT, Hoh BL, Janis LS, Kase CS, Kleindorfer DO, Lee JM, Moseley ME, Peterson ED, Turan TN, Valderrama AL, Vinters HV; American Heart Association Stroke Council, Council on Cardiovascular Surgery and Anesthesia; Council on Cardiovascular Radiology and Intervention; Council on Cardiovascular and Stroke Nursing; Council on Epidemiology and Prevention; Council on Peripheral Vascular Disease; Council on Nutrition, Physical Activity and Metabolism. An updated definition of stroke for the 21st century: a statement for healthcare professionals from the American Heart Association/American Stroke Association. Stroke. 2013 Jul;44(7):2064-89. doi: 10.1161/STR.0b013e318296aeca. Epub 2013 May 7. PMID 23652265
- [Background] Einstein AJ, Henzlova MJ, Rajagopalan S. Estimating risk of cancer associated with radiation exposure from 64-slice computed tomography coronary angiography. JAMA. 2007 Jul 18;298(3):317-23. doi: 10.1001/jama.298.3.317. PMID 17635892
- [Background] Barrett BJ, Katzberg RW, Thomsen HS, Chen N, Sahani D, Soulez G, Heiken JP, Lepanto L, Ni ZH, Ni ZH, Nelson R. Contrast-induced nephropathy in patients with chronic kidney disease undergoing computed tomography: a double-blind comparison of iodixanol and iopamidol. Invest Radiol. 2006 Nov;41(11):815-21. doi: 10.1097/01.rli.0000242807.01818.24. PMID 17035872
- [Derived] Whittington B, Tzolos E, Bing R, Andrews J, Lucatelli C, MacAskill MG, Tavares AAS, Clark T, Mills NL, Nash J, Dey D, Slomka PJ, Koglin N, Stephens AW, van Beek EJR, Smith C, Dweck MR, Williams MC, Whiteley W, Wardlaw JM, Newby DE. Noninvasive In Vivo Thrombus Imaging in Patients With Ischemic Stroke or Transient Ischemic Attack-Brief Report. Arterioscler Thromb Vasc Biol. 2023 Sep;43(9):1729-1736. doi: 10.1161/ATVBAHA.122.318204. Epub 2023 Jul 13. PMID 37439259
- [Derived] Tzolos E, Bing R, Andrews J, MacAskill MG, Tavares AAS, Macnaught G, Clark T, Mills NL, Fujisawa T, Nash J, Dey D, Slomka PJ, Koglin N, Stephens AW, Deutsch MA, van Beek EJR, Williams MC, Hermann S, Hugenberg V, Dweck MR, Newby DE. Noninvasive In Vivo Coronary Artery Thrombus Imaging. JACC Cardiovasc Imaging. 2023 Jun;16(6):820-832. doi: 10.1016/j.jcmg.2022.10.002. Epub 2022 Dec 14. PMID 36526577
- See also: Related Info — https://www.edinburghcrf.ed.ac.uk/